CLINICAL TRIAL: NCT05879705
Title: The Effectiveness of OT-ParentShip on Parental Resilience and Functioning of Adolescents With High Functioning Autism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0119-20-COM
Record Dates: First submitted 2023-03-20; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; RCT; Parent-intervention; Adolescents
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: A mixed method, two group, randomized controlled trial (RCT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- An OT-ParentShip intervention (Experimental): Each family will participate in a series of 11 individual weekly sessions of 90 minutes each and another session after three months from the end of the intervention.
  Interventions: Other: Parent intervention
- A psycho-educational intervention group. (Other): Each family will receive a general, psycho-educational, video-based intervention. The program includes 6 videos with an average length of 20 minutes each.The participants are asked to watch the video according to the order once every two weeks.
  Interventions: Other: Parent intervention

INTERVENTIONS:
Other: Parent intervention — Family centered, strength-based, Occupational therapy intervention program

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of the OT (Occupational Therapy)-ParentShip intervention program for parents of adolescents with Autism. A mixed method, two group, randomized controlled trial (RCT). Forty participants will be recruited through convenience sampling and will be randomly assigned to one of two groups: an OT-ParentShip intervention group or a psycho-educational intervention group.

The main questions it aims to answer are:

* Which baseline characteristics will predict positive treatment outcomes (based on the outcome measures defined)?
* What is the parents' perception and experience from the intervention process and its outcomes?

The course of intervention in each group:

OT-ParentShip group: each family will participate in a series of 11 individual weekly sessions of 90 minutes each and another session after three months from the end of the intervention. Control group: Each family will receive a general, psycho-educational, video-based intervention.

DETAILED DESCRIPTION:
Parents of adolescents with Autism Spectrum Disorder (ASD) are at risk for low parental competence and decreased sense of autonomy, facing challenges in parent-child relationships. Moreover, parents of children with High Functioning ASD (HFASD) experience significantly higher levels of parental stress in comparison to parents of typically developing children. A range of body functions is associated with occupational challenges in ASD, such as sensory, cognitive, social-communicative and emotional. Occupation based interventions consistent with Self-Determination Theory (SDT) principles were found to promote parental competence and improve participation of children with ASD. However, there is a need for multidimensional interventions that address both the adolescents' occupational challenges and underlying body functions, as well as parents' psychological needs. OT (Occupational Therapy)-ParentShip is an intervention program for parents of adolescents with HFASD which includes an integrative multidimensional approach to the multiple factors involved in the functioning of adolescents with HFASD and aims to promote parental resilience and enhance adolescents' participation.

Preliminary results: a mixed methods pilot study (N=10) was conducted to evaluate the feasibility of the OT-ParentShip. Significant improvements were found in parents' and adolescents' functional goals, as well as improvement in parental resilience. In addition, six themes were identified, shedding light on the therapeutic components and change mechanisms of OT-Parentship.

ELIGIBILITY:
Inclusion Criteria:

Phase A:

* Parents (father, mother or both) of an adolescent (male or female) aged 12- 18, who is a student in junior or high school.
* Medical diagnosis (by a neurologist or psychiatrist) of a HFASD (Level 1) according to the criteria of DSM-5 or DSM-IV.
* Parents report regarding unmet functional needs / difficulties.
* Signed consent of at least one parent to attend all sessions for a period of approximately 13 weeks.

Phase B:

• Receiving a score that defines disability in at least one of the following areas: sensory processing / executive function / social-communication skills.

Exclusion Criteria:

* Unbalanced neurologic or psychiatric comorbidity with HFASD, having a major effect on functioning, based on parental report.
* Parents who are unable or unavailable (emotionally or for any other reason) to participate in the intervention or the implementation (based on self-report).

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Autism: Parenting Questionnaire (APQ) (Kim, Anderson, Birkin, Seymour, & Moore, 2004). | Before intervention (Time 1)
  A self-completed questionnaire which surveys parents on six domains of autism-specific parenting competence (knowledge, communication, play, behavior management, security and family functioning) and one domain of parenting stress.
Basic Psychological Need Satisfaction in Relationships (La Guardia, Ryan, Couchman, & Deci 2000). | Before intervention (Time 1)
  This questionnaire used in order to assess the degree to which a person experiences basic need satisfaction while relating to his or her spouse, best friend, mother, children, or whomever.
Canadian Occupational Performance Measure (COPM)- Parent (Law, Baptiste, Carswell, McColl, Polatajko, & Pollock, 1998) | Before intervention (Time 1)
  A semi-structured interview, used as an outcome measure to detect changes in self-perception of patient performance and satisfaction over time by identifying problems with daily functioning.
Autism: Parenting Questionnaire (APQ) (Kim, Anderson, Birkin, Seymour, & Moore, 2004). | Immediately post intervention (Time 2)
  A self-completed questionnaire which surveys parents on six domains of autism-specific parenting competence (knowledge, communication, play, behavior management, security and family functioning) and one domain of parenting stress.
Basic Psychological Need Satisfaction in Relationships (La Guardia, Ryan, Couchman, & Deci 2000). | Immediately post intervention (Time 2)
  This questionnaire used in order to assess the degree to which a person experiences basic need satisfaction while relating to his or her spouse, best friend, mother, children, or whomever.
Canadian Occupational Performance Measure (COPM)- Parent (Law, Baptiste, Carswell, McColl, Polatajko, & Pollock, 1998) | Immediately post intervention (Time 2)
  A semi-structured interview, used as an outcome measure to detect changes in self-perception of patient performance and satisfaction over time by identifying problems with daily functioning.
Autism: Parenting Questionnaire (APQ) (Kim, Anderson, Birkin, Seymour, & Moore, 2004). | Three months post intervention (follow-up-Time 3).
  A self-completed questionnaire which surveys parents on six domains of autism-specific parenting competence (knowledge, communication, play, behavior management, security and family functioning) and one domain of parenting stress.
Basic Psychological Need Satisfaction in Relationships (La Guardia, Ryan, Couchman, & Deci 2000). | Three months post intervention (follow-up-Time 3).
  This questionnaire used in order to assess the degree to which a person experiences basic need satisfaction while relating to his or her spouse, best friend, mother, children, or whomever.
Canadian Occupational Performance Measure (COPM)- Parent (Law, Baptiste, Carswell, McColl, Polatajko, & Pollock, 1998) | Three months post intervention (follow-up-Time 3).
  A semi-structured interview, used as an outcome measure to detect changes in self-perception of patient performance and satisfaction over time by identifying problems with daily functioning.
Canadian Occupational Performance Measure (COPM)- Parent (Law, Baptiste, Carswell, McColl, Polatajko, & Pollock, 1998)- Transfer goal | Immediately post intervention
  A semi-structured interview, used as an outcome measure to detect changes in self-perception of patient performance and satisfaction over time by identifying problems with daily functioning.
Canadian Occupational Performance Measure (COPM)- Parent (Law, Baptiste, Carswell, McColl, Polatajko, & Pollock, 1998)- Transfer goal | Three months post intervention
  A semi-structured interview, used as an outcome measure to detect changes in self-perception of patient performance and satisfaction over time by identifying problems with daily functioning.

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure (COPM)-Adolescent (Law, Baptiste, Carswell, McColl, Polatajko, & Pollock, 1998) | Before intervention (Time 1)
  A semi-structured interview, used as an outcome measure to detect changes in self-perception of patient performance and satisfaction over time by identifying problems with daily functioning.
Canadian Occupational Performance Measure (COPM)-Adolescent (Law, Baptiste, Carswell, McColl, Polatajko, & Pollock, 1998) | Immediately post intervention (Time 2)
  A semi-structured interview, used as an outcome measure to detect changes in self-perception of patient performance and satisfaction over time by identifying problems with daily functioning.
Canadian Occupational Performance Measure (COPM)-Adolescent (Law, Baptiste, Carswell, McColl, Polatajko, & Pollock, 1998) | Three months post intervention (follow-up-Time 3)
  A semi-structured interview, used as an outcome measure to detect changes in self-perception of patient performance and satisfaction over time by identifying problems with daily functioning.
Canadian Occupational Performance Measure (COPM)-Adolescent (Law, Baptiste, Carswell, McColl, Polatajko, & Pollock, 1998)- Transfer goal | Immediately post intervention
  A semi-structured interview, used as an outcome measure to detect changes in self-perception of patient performance and satisfaction over time by identifying problems with daily functioning.
Canadian Occupational Performance Measure (COPM)-Adolescent (Law, Baptiste, Carswell, McColl, Polatajko, & Pollock, 1998)- Transfer goal | Three months post intervention
  A semi-structured interview, used as an outcome measure to detect changes in self-perception of patient performance and satisfaction over time by identifying problems with daily functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Batel Wachspress, MA, Study Director — Hebrew University of Jerusalem
Locations (1):
- The Hebrew University of Jerusalem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wachspress B, Maeir A, Mazor-Karsenty T. Content Validity of the Parentship Protocol: A Multidimensional Intervention for Parents of Adolescents with High-Functioning Autism Spectrum Disorder. Phys Occup Ther Pediatr. 2019;39(4):373-387. doi: 10.1080/01942638.2018.1500968. Epub 2018 Sep 6. PMID 30188233